CLINICAL TRIAL: NCT05670288
Title: Impact of Gut Microbiome on Metabolic and Bowel Function During the First Year After Spinal Cord Injury
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Pittsburgh Medical Center (Other); Craig Hospital (Other); Rancho Los Amigos National Rehabilitation Center (Other)
Responsible Party: Principal Investigator, Jereme Wilroy, Associate Professor, University of Alabama at Birmingham
Other Study IDs: IRB-300010011; 90SIMS0020 (Other Grant/Funding Number: National Institute on Disability, Independent Living, and Rehabilitation Research)
Record Dates: First submitted 2022-12-08; First posted 2023-01-04 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries; Gut Microbiome
Keywords: SCI; Inflammation; Bowel Function; Blood Sugar; Lipid Profiles
MeSH Terms: conditions — Spinal Cord Injuries; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool and Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spinal Cord Injury: Patients who have had an acute spinal cord injury in the past 72 hours

SUMMARY:
The Investigators will recruit 35 participants with acute SCI (within 6 weeks of injury) Fasting blood collection and bowel function survey will be conducted 3 times: at baseline [within 6 weeks of injury], 6, and 12 months after SCI. Stool will be collected for gut microbiome analysis 3 times.

DETAILED DESCRIPTION:
Stool and fasting blood collection will occur at the rehabilitation hospital (during in-patient stay) and at participants' homes. During the hospital stay, stool will be collected at the bedside by the research team and placed in a Para-pak® vial for sample preservation. Blood will also be collected by the research team.

For sample collection at home, a research nurse will travel to participants home to perform blood draws and bing back to the research lab for processing/analysis/storage.

The nurse may also collect the stool sample at the same time as the blood draw if available. If not, participants and their caregivers will be provided with a pre-paid/labeled FedEx package containing a stool collection kit (Para-pak® vial). Prior to bowel movement, participants and caregivers will be asked to clean the anal area using the sanitizing wipes; approximately 5-10 mL of stool will be transferred to the Para-pak® vial using the attached spatula in the Para-pak® vial. For participants who conduct their bowel management program in their beds, an additional sterile absorbent pad will be provided to use as a barrier between the bed and the participant to limit contamination. FedEx package containing the stool sample will be shipped to the investigators' lab

For each participant, the Investigators will record 1) diet (via 24-hour dietary recalls), 2) physical activity habits (via the rehabilitation therapies survey included in the SCI common data elements [CDEs], 3)Leisure Time Physical Activity Questionnaire; 4)depression and anxiety (via Patient Health Questionnaire-9 [PHQ9] and the General Anxiety Disorder-7 scale (GAD7),respectively); 5)prescribed medications, including antibiotics (via RedCap platform); 6)use of supplements and bowel routine components, including probiotics and laxatives (via self-report); and 7)any other comorbidities beyond GI dysfunction

ELIGIBILITY:
Inclusion Criteria:

1. 18-85 years of age
2. diagnosis of traumatic SCI at the cervical to lumbar level (C3-L2)
3. classification of A, B, C (motor complete, incomplete).

Exclusion Criteria:

1. Women who are pregnant prior to consent
2. neurological impairment other than SCI
3. self-reported history of Crohn's disease or diverticulitis
4. irritable bowel syndrome
5. gastric blockage/obstruction or swallowing disorder
6. prior GI surgery
7. intrathecal pump
8. concurrent usage of functional electrical stimulation for bowel management (e.g., constipation).
9. able to ambulate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had an acute spinal cord injury in the past 6 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Neurological impairment - Injury level by ISNCSCI | Baseline
  Injury level determined by International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) exam
Neurological impairment - Injury level by AIS | Baseline
  Injury level determined by American Spinal Injury Association Impairment Scale (AIS). classification.
Neurological impairment - completeness of injury by ISNCSCI | Baseline
  Completeness of injury determined by International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) exam
Neurological impairment - completeness of injury by AIS | Baseline
  Completeness of injury determined by American Spinal Injury Association Impairment Scale (AIS). classification.
Neurological impairment - Injury level by ISNCSCI | Month 6
  Injury level determined by International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) exam
Neurological impairment - Injury level by AIS | Month 6
  Injury level determined by American Spinal Injury Association Impairment Scale (AIS). classification.
Neurological impairment - completeness of injury by ISNCSCI | Month 6
  Completeness of injury determined by International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) exam
Neurological impairment - completeness of injury by AIS | Month 6
  Completeness of injury determined by American Spinal Injury Association Impairment Scale (AIS). classification.
Neurological impairment - Injury level by ISNCSCI | Month 12
  Injury level determined by International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) exam
Neurological impairment - Injury level by AIS | Month 12
  Injury level determined by American Spinal Injury Association Impairment Scale (AIS). classification.
Neurological impairment - completeness of injury by ISNCSCI | Month 12
  Completeness of injury determined by International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) exam
Neurological impairment - completeness of injury by AIS | Month 12
  Completeness of injury determined by American Spinal Injury Association Impairment Scale (AIS). classification.
Microbiome composition - Bacterial 16S rRNA sequincing | Baseline
  Bacterial 16S rRNA sequencing will be performed
Microbiome composition - Bacterial 16S rRNA sequincing | Month 1
  Bacterial 16S rRNA sequencing will be performed
Microbiome composition - Bacterial 16S rRNA sequincing | Month 6
  Bacterial 16S rRNA sequencing will be performed
Microbiome composition - Bacterial 16S rRNA sequincing | Month 12
  Bacterial 16S rRNA sequencing will be performed
Microbiome composition - Metagenomics | Baseline
  A subset of 16S rRNA gene surveys that show differences in taxa and alpha and beta diversity are selected for follow-up via shotgun metagenomics.
Microbiome composition - Metagenomics | Month 1
  A subset of 16S rRNA gene surveys that show differences in taxa and alpha and beta diversity are selected for follow-up via shotgun metagenomics.
Microbiome composition - Metagenomics | Month 6
  A subset of 16S rRNA gene surveys that show differences in taxa and alpha and beta diversity are selected for follow-up via shotgun metagenomics.
Microbiome composition - Metagenomics | Month 12
  A subset of 16S rRNA gene surveys that show differences in taxa and alpha and beta diversity are selected for follow-up via shotgun metagenomics.
Gut derived metabolites | Baseline
  Blood will be collected and serum extract metabolites will be isolated
Gut derived metabolites | Month 1
  Blood will be collected and serum extract metabolites will be isolated
Gut derived metabolites | Month 6
  Blood will be collected and serum extract metabolites will be isolated
Gut derived metabolites | Month 12
  Blood will be collected and serum extract metabolites will be isolated
Analysis of metabolic markers to determine metabolic function | Baseline
  Blood will be collected and serum assays for metabolic markers performed
Analysis of metabolic markers to determine metabolic function | Month 1
  Blood will be collected and serum assays for metabolic markers performed
Analysis of metabolic markers to determine metabolic function | Month 6
  Blood will be collected and serum assays for metabolic markers performed
Analysis of metabolic markers to determine metabolic function | Month 12
  Blood will be collected and serum assays for metabolic markers performed
Analysis of inflammatory markers to determine Inflammatory state | Baseline
  Blood will be collected and serum assays for inflammatory markers performed
Analysis of inflammatory markers to determine Inflammatory state | Month 1
  Blood will be collected and serum assays for inflammatory markers performed
Analysis of inflammatory markers to determine Inflammatory state | Month 6
  Blood will be collected and serum assays for inflammatory markers performed
Analysis of inflammatory markers to determine Inflammatory state | Month 12
  Blood will be collected and serum assays for inflammatory markers performed
Bowel function - International Bowel Function Basic and Extended Data Set Assessment | Baseline
  International Bowel Function Basic and Extended Data Set assessment will be utilized to assess bowel-related symptoms.
Bowel function - Bristol Stool Scale | Baseline
  Bristol Stool Scale assessment will be utilized to assess bowel-related symptoms.
Bowel function - International Bowel Function Basic and Extended Data Set Assessment | Month 1
  International Bowel Function Basic and Extended Data Set assessment will be utilized to assess bowel-related symptoms.
Bowel function - Bristol Stool Scale | Month 1
  Bristol Stool Scale assessment will be utilized to assess bowel-related symptoms.
Bowel function - International Bowel Function Basic and Extended Data Set Assessment | Month 6
  International Bowel Function Basic and Extended Data Set assessment will be utilized to assess bowel-related symptoms.
Bowel function - Bristol Stool Scale | Month 6
  Bristol Stool Scale assessment will be utilized to assess bowel-related symptoms.
Bowel function - International Bowel Function Basic and Extended Data Set Assessment | Month 12
  International Bowel Function Basic and Extended Data Set assessment will be utilized to assess bowel-related symptoms.
Bowel function - Bristol Stool Scale | Month 12
  Bristol Stool Scale assessment will be utilized to assess bowel-related symptoms.

SECONDARY OUTCOMES:
Diet | Baseline
  Participant records 24-hour dietary recalls
Diet | Month 1
  Participant records 24-hour dietary recalls
Diet | Month 6
  Participant records 24-hour dietary recalls
Diet | Month 12
  Participant records 24-hour dietary recalls
Physical activity - PARA-SCI | Baseline
  Complete PARA-SCI questionnaire to determine physical activity level
Physical activity - CDEs | Baseline
  Complete rehabilitation therapies survey (CDEs) to determine physical activity level
Physical activity - PARA-SCI | Month 1
  Complete PARA-SCI questionnaire to determine physical activity level
Physical activity - CDEs | Month 1
  Complete rehabilitation therapies survey (CDEs) to determine physical activity level
Physical activity - PARA-SCI | Month 6
  Complete PARA-SCI questionnaire to determine physical activity level
Physical activity - CDEs | Month 6
  Complete rehabilitation therapies survey (CDEs) to determine physical activity level
Physical activity - PARA-SCI | Month 12
  Complete PARA-SCI questionnaire to determine physical activity level
Physical activity - CDEs | Month 12
  Complete rehabilitation therapies survey (CDEs) to determine physical activity level
Medication List - Medical Record Review | Baseline
  Medical record review of prescribed medications being taken
Medication List - Self-report | Baseline
  Self-report of prescribed medications being taken
Medication List - Medical Record Review | Month 1
  Medical record review of prescribed medications being taken
Medication List - Self-report | Month 1
  Self-report of prescribed medications being taken
Medication List - Medical Record Review | Month 6
  Medical record review of prescribed medications being taken
Medication List - Self-report | Month 6
  Self-report of prescribed medications being taken
Medication List - Medical Record Review | Month 12
  Medical record review of prescribed medications being taken
Medication List - Self-report | Month 12
  Self-report of prescribed medications being taken
Supplement usage - Medical Record Review | Baseline
  Medical record review of supplements being taken
Supplement usage - self-report | Baseline
  Self-report of supplements being taken
Supplement usage - Medical Record Review | Month 1
  Medical record review of supplements being taken
Supplement usage - self-report | Month 1
  Self-report of supplements being taken
Supplement usage - Medical Record Review | Month 6
  Medical record review of supplements being taken
Supplement usage - self-report | Month 6
  Self-report of supplements being taken
Supplement usage - Medical Record Review | Month 12
  Medical record review of supplements being taken
Supplement usage - self-report | Month 12
  Self-report of supplements being taken
Depression | Baseline
  Complete PHQ9 questionnaires to determine depression level
Depression | Month 1
  Complete PHQ9 questionnaires to determine depression level
Depression | Month 6
  Complete PHQ9 questionnaires to determine depression level
Depression | Month 12
  Complete PHQ9 questionnaires to determine depression level
Anxiety | Baseline
  Complete GAD7 questionnaire to determine anxiety level
Anxiety | Month 1
  Complete GAD7 questionnaire to determine anxiety level
Anxiety | Month 6
  Complete GAD7 questionnaire to determine anxiety level
Anxiety | Month 12
  Complete GAD7 questionnaire to determine anxiety level
Comorbidities | Baseline
  Evaluate Medical history (CDEs) for any other comorbidities beyond GI dysfunction
Comorbidities | Month 1
  Evaluate Medical history (CDEs) for any other comorbidities beyond GI dysfunction
Comorbidities | Month 6
  Evaluate Medical history (CDEs) for any other comorbidities beyond GI dysfunction
Comorbidities | Month 12
  Evaluate Medical history (CDEs) for any other comorbidities beyond GI dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Jereme Wilroy, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingahm, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No